CLINICAL TRIAL: NCT06855433
Title: A Randomized, Double-Blind, Multi-Site Placebo Controlled Trial of Colchicine in Calcium Pyrophosphate Deposition Disease
Brief Title: Colchicine to Reduce Your SympToms And Lower Levels of Inflammation, Zeroing in on Effective CPPD Disease Treatment
Acronym: CRYSTALLIZE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Rheumatology Research Foundation (Other)
Responsible Party: Principal Investigator, Sara Tedeschi, M.D., M.P.H., Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024P003512
Record Dates: First submitted 2025-02-26; First posted 2025-03-03 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: CPPD - Calcium Pyrophosphate Deposition Disease
Keywords: colchicine; CPPD disease; calcium pyrophosphate; pseudogout
MeSH Terms: conditions — Chondrocalcinosis | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data Coordinating Center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Colchicine (Experimental): Colchicine
  Interventions: Drug: Colchicine Pill
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine Pill — Colchicine 0.6mg tab, overencapsulated to match placebo capsule, taken by mouth once daily
  Arms: Colchicine
Drug: Placebo — Placebo capsule, taken by mouth once daily
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if colchicine reduces levels of proteins indicating inflammation in the blood in individuals with calcium pyrophosphate deposition (CPPD) disease. The trial will also test the effect of colchicine on joint symptoms in CPPD disease. The main questions it aims to answer are:

* Does colchicine reduce the level of interleukin 18 (IL-18) in the blood of individuals with CPPD disease?
* Does colchicine reduce pain scores in individuals with CPPD disease?

Researchers will compare colchicine once daily to a placebo (a look-alike pill that contains no drug) to see if colchicine works to treat CPPD disease.

Participants will:

* Take colchicine or a placebo every day for 6 months
* Visit the clinic 3 times in 6 months for joint examinations, surveys, and blood tests. Each visit will last 2-3 hours.
* Speak on the telephone with researchers for about 4 times over 6 months. Each phone call will last about 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Fulfill ACR/EULAR 2023 CPPD classification criteria
* Acute or chronic joint inflammation in the past 3 months, not attributable to another condition
* Pain visual analog scale (pain VAS) >=30 at screening

Exclusion Criteria:

* age <40 years
* chronic diarrhea
* gout, rheumatoid arthritis, or psoriatic arthritis
* cirrhosis
* ongoing use of colchicine and unwilling to undergo a 30-day wash-out period (note: patients using colchicine at screening can enroll if they agree to a 30-day wash-out before randomization)
* pregnant or breast-feeding
* use of methotrexate, hydroxychloroquine, or anakinra in the past month
* use of oral glucocorticoid in the past week
* use of strong CYP3A4 inhibitors per FDA package insert for colchicine
* use of P-glycoprotein inhibitors per FDA package insert for colchicine
* known allergy to colchicine

Screening labs with any of the following:

* hemoglobin < 11.5 g/dL
* WBC <3 x 10^9/L
* platelets <110 x10^9/L
* creatinine clearance (CrCl) <30 mL/min
* ALT or AST >3x upper limit of normal (ULN)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-04-10 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Interleukin 18 (IL-18) | Baseline and Week 24
  Serum IL-18

SECONDARY OUTCOMES:
Serum IL-1b | Baseline and Week 24
  Serum IL-1b
Serum IL-17A | Baseline and Week 24
  Serum IL-17A
High-sensitivity C-reactive protein (hsCRP) | Baseline and Week 24
  High-sensitivity C-reactive protein in blood
IL-1b gene signature expression in PBMCs | Baseline and Week 24
  Expression of a panel of genes involved in IL-1b production or signaling, as percentage of total gene expression per cell
Immune cell population frequencies | Baseline and Week 24
  Immune cell clusters among PBMCs
Pain visual analog scale (pain VAS) | Baseline, Week 12, Week 24
  Pain VAS (range 0-100mm) reflecting pain in the past 24 hours due to CPPD disease
Patient Reported Outcome Measurement Information System (PROMIS)-Pain Interference | Baseline, Week 12, Week 24
  PROMIS-Pain Interference Short Form 6b, assessing pain interference in the past 7 days. (T-score range 0-100, with higher scores indicating greater pain interference)
Patient Reported Outcome Measurement Information System (PROMIS)-Physical Function | Baseline, Week 12, Week 24
  PROMIS-Physical Function Short Form 10a (T-score range 0-100, with higher scores indicating better physical function)
Patient Global Assessment of Response to Treatment | Week 12, Week 24
  5 point Likert scale
Patient Global Assessment | Baseline, Week 12, Week 24
  Patient Global Assessment of CPPD Disease Activity (range: 0-10)
Assessor Global Assessment | Baseline, Week 12, Week 24
  Assessor's Global Assessment of CPPD Disease Activity (range: 0-10)
Flare count | Week 12, Week 24
  Number of acute calcium pyrophosphate crystal arthritis flares
Adverse events | Week 12, Week 24
  Number of expected adverse events and unexpected adverse events